CLINICAL TRIAL: NCT00823004
Title: GnRH Antagonist /Letrozole Versus Microdose GnRH Agonist Flare Protocol in Poor Responders Undergoing in Vitro Fertilization
Brief Title: Antagonist/Letrozole in Poor Responders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: Principal Investigator, homa oskouian, fellowship, Yazd Research & Clinical Center for Infertility
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1969yazdRCCI
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Ovarian Stimulation
Keywords: controlled ovarian hyperstimulation; pregnancy rate; Poor responders; GnRH antagonist; GnRH agonist; letrozole; in vitro fertilization
MeSH Terms: interventions — Letrozole; lactitol; Contraceptives, Oral; Desogestrel; Gonadotropin-Releasing Hormone; Buserelin; follitropin alfa; hMG-IBSA; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): A/L: Poor responders who will receive letrozole and GnRH antagonist for ovarian stimulation
  Interventions: Drug: letrozole; Drug: oral contraceptive (Marvelone); Drug: recombinant FSH or hMG; Drug: ganirelix acetate
- 2 (Active Comparator): MF: In this arm poor responders are treated by microdose GnRH agonist flare protocol
  Interventions: Drug: oral contraceptive (Marvelone); Drug: GnRH agonist (buserelin); Drug: recombinant FSH or hMG

INTERVENTIONS:
Drug: letrozole — letrozole 5mg/day from day 3 to day 7 of menstrual cycle
  Other Names: letrozole (Femara, Novartis, East Hanover, NJ)
  Arms: 1
Drug: oral contraceptive (Marvelone) — oral contraceptive, first 21 days
  Other Names: Marvelon
Drug: GnRH agonist (buserelin) — 50 µg SC twice daily
  Other Names: suprefact
  Arms: 2
Drug: recombinant FSH or hMG — recombinant FSH or hMG 300-450 IU/day
  Other Names: Gonal F; Merional
Drug: ganirelix acetate — GnRH antagonist (ganirelix acetate) when a leading follicle reaches a mean diameter of 14 mm, 0.25 mg per day (Antagon, Organon, West Orange, NJ)
  Other Names: Antagon
  Arms: 1

SUMMARY:
Failure to respond to controlled ovarian hyperstimulation (COH) is still a major concern in assisted reproduction and there is no consensus on the ovarian stimulation choice regime for poor responders.

Aim: To evaluate and compare the efficacy of a microdose GnRH agonist flare (MF) and a GnRH antagonist/letrozole (A/L) protocols in poor responders undergoing in vitro fertilization (IVF).

Methods: One hundred eighty poor responder patients will be randomized to an ovarian stimulation protocol with either a MF or a letrozole and high dose FSH/hMG and flexible GnRH antagonist protocol.

DETAILED DESCRIPTION:
All women receive 21 days of an oral contraceptive. A MF protocol will be used for ovarian stimulation in 90 patients. Three days after the last pill, a GnRH-agonist buserelin (Suprefact, Aventis Pharma, Frankfurt, Germany) 50 µg SC twice daily will be initiated and two days after that, recombinant FSH (Gonal-F, Serono, Aubonne, Switzerland) or hMG (Merional, IBSA, Lugano, Switzerland) 300-450 IU/day will be administered. Ninetyty patients will be assigned to an A/L protocol. After oral contraceptive withdrawal bleeding on day 3 of cycle, recombinant FSH or hMG 300-450 IU/day will be initiated and letrozole (Femara, Novartis, East Hanover, NJ) 5 mg/day will be administered for 5 days. When the dominant follicle reached 14 mm in mean diameter, ganirelix acetate (Antagon, Organon, West Orange, NJ) 0.25 mg SC daily will be started.

Patients weill be monitored by serial vaginal ultrasonography and measurement of serum E2 level. When at least two follicles with a mean diameter of 18 mm will be achieved hCG (Pregnyl, Organon, Oss, the Netherlands) 10000 IU will be administered. Cycle cancellation will be considered when fewer than two follicles with normal growth pattern weill be noted.

Oocyte retrieval will be performed 34-36 hours after hCG administration. Conventional IVF or intracytoplasmic sperm injection (ICSI) will be performed as appropriate. Embryos with 4-6 equally sized blastomers on day 2 with ≤ 20% fragmentation and no multinucleation will be considered top quality embryos. Embryos with 2-6 equally or unequally blastomers with ≤20% fragmentation and no multinucleation will be considered good quality embryos. Embryos will be transferred on day 2 or 3 under ultrasound guidance, with a C.C.D. embryo transfer catheter ( Laboratoire C.C.D., Paris, France). Luteal support with progesterone in oil (Progesterone, Aburaihan Co., Tehran, Iran) 100 mg daily IM will be started on the day of oocyte retrieval.

Serum β-hCG level will be measured 14 days after embryo transfer and a transvaginal ultrasonography will be performed 3 weeks after positive β-hCG for documentation of gestational sac and fetal heart activity. Clinical pregnancy will be considered as the presence of a gestational sac with fetal heart activity.

ELIGIBILITY:
Inclusion Criteria:

* at least one previous failed IVF cycle in which three or fewer follicles with a mean diameter of 16 mm were achieved, and/or
* serum E2 level measured on the day of hCG administration was ≤500 pg/ml

Exclusion Criteria:

* day 3 serum FSH level ≥12 mIU/mL
* there is no age limit

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 5 weeks

SECONDARY OUTCOMES:
stimulation outcomes | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: homa oskouian, M.D., Principal Investigator — Research and clinical center for infertility; robab davar, MD, Principal Investigator — Research and clinical center for infertility
Locations (1):
- Research and clinical center for infertility, Yazd, Yazd Province, Iran